CLINICAL TRIAL: NCT00869167
Title: Ramelteon for Insomnia Comorbid With Asthma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Brandon Lu, Physician, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-052R
Record Dates: First submitted 2009-03-19; First posted 2009-03-25 (Estimated); Results first posted 2012-06-29 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Insomnia; Asthma
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Asthma | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Ramelteon (Experimental)
  Interventions: Drug: Ramelteon
- 2: Placebo (Placebo Comparator)
  Interventions: Drug: Ramelteon

INTERVENTIONS:
Drug: Ramelteon — melatonin agonist
  Other Names: Rozerem

SUMMARY:
This trial will test the efficacy and safety of ramelteon, a selective melatonin agonist, on patients with insomnia comorbid with asthma.

DETAILED DESCRIPTION:
Subjects with insomnia comorbid with asthma will be randomized to placebo or ramelteon at night for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 60 with both insomnia and asthma.
* Insomnia:

  * a complaint of difficulty initiating sleep, difficulty maintaining sleep, or waking up too early or sleep that is chronically nonrestorative or poor in quality,
  * the sleep difficulty occurs despite adequate opportunity and circumstances for sleep, and
  * at least one form of daytime impairment related to the nighttime sleep difficulty must be present. The sleep complaint should be present on most days for at least 3 months.
* Additional inclusion criteria include: a subjective TST <6.5 h and a subjective SL > 45 min per night; a mean LPS >20 min over 2 consecutive nights by polysomnography (neither night could have been <15 min); a habitual bedtime between 10 PM and 1 AM; and ISI score > 10 (based on 0-4 scale). LPS is defined as amount of time to the first 10 minutes of continuous sleep.
* Asthma will be diagnosed based on suggestive clinical history and either

  * airway hyperresponsiveness indicated by a 20% or greater decrease in FEV1 in response to inhalation of methacholine at 8 mg/mL or less
  * bronchodilator-responsive expiratory airflow limitation (if FEV1 < 70% of predicted value or < 1.5 L, improving ≥200 mL and 12% in response to 180 µg of albuterol aerosol). In addition to the above criteria, patients should have well-controlled asthma as evidenced by ACQ score < 1.5.

Exclusion Criteria:

* Primary sleep pathology, other than insomnia as assessed by sleep history and confirmed by polysomnography to exclude significant sleep apnea (RDI > 15), periodic leg movements (movement arousal index > 15), REM behavior disorder; or circadian sleep-wake disorders
* History of cognitive or other neurological disorders;
* History of DSM-IV criteria for any major psychiatric disorder, including mania or alcohol or substance abuse;
* Depressive symptoms as assessed by the CES-D. Subjects with a score of 22 or greater indicates that the person may be suffering from a major depression and therefore, will be referred to their physician;
* Unstable or serious medical conditions;
* Current, or use within the past month, of psychoactive, hypnotic, stimulant or analgesic medications (except occasionally);
* Shift work or other types of self imposed irregular sleep schedules;
* Obesity (BMI > 35 Kg/m2); or
* Pregnancy or desire to become pregnant during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon S Lu, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ramelteon; Placebo: Participants with insomnia and asthma are randomized to Ramelteon 8mg and sleep hygiene for 5 weeks or to placebo and sleep hygiene for 5 weeks. Ramelteon or placebo to be taken within 30 minutes before
Period: Overall Study
Arm/Group | Ramelteon | Placebo
Started | 2 | 1
Completed | 2 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramelteon | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.5 (9.2) | 38 | 35.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Sleep Quality Index
Description: The change in ISI and PSQI from baseline to end of study will be compared between the two groups.
  PSQI has a score range of 0-21, with lower the number being less sleep disturbances ISI has a score range of 0-28, with lower score meaning less insomnia symptoms
Time Frame: baseline and post-treatment (at end of 5 weeks)
Population: The 2 subjects in the Ramelteon group completed the study. The 1 subject in the placebo group did not complete the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 2 | 0
units on a scale | 2 (0) |

2. Secondary Outcome: Daytime Sleepiness (Epworth Sleepiness Scale)
Description: Score of 0-24, with 24 being the most sleepy
Time Frame: baseline and post-treatment (at end of 5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 2 | 0
units on a scale | 3.5 (0.7) |

3. Secondary Outcome: Daytime Performance (Digit Symbol Substitution Test)
Description: DSST tests the number of correct digit-symbol pairs that an individual can identify within an allotted period (60-90 sec). It test memory and concentration, among other parameters.
  DSST score can range from 0-125, with 125 being the most number correct during the allotted time period.
Time Frame: baseline and post-treatment (at end of 5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number correct
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 2 | 0
Number correct | 8 (1.4) |

4. Secondary Outcome: Daytime Lung Function (Peak Flow Monitoring) in Liter/Min
Time Frame: baseline and during treatment period (during 5th week)
Population: This measure was added during the study and no subjects completed the measure.
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Insomnia Severity Index
Description: as for outcome 1
Time Frame: 5 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ramelteon; Placebo: Participants with insomnia and asthma are randomized to Ramelteon 8mg and sleep hygiene for 5 weeks or to placebo and sleep hygiene for 5 weeks. Ramelteon or placebo to be taken within 30 minutes before bedtime
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 2 | 0
units on a scale | -6.5 (6.36) |

ADVERSE EVENTS:
Arm/Group | Ramelteon | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

LIMITATIONS AND CAVEATS:
Recruitment difficulties led to only 3 participants in the study. Only 2 participants finished the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No